CLINICAL TRIAL: NCT01955265
Title: Promoting Adolescent Development Through Sports in Hong Kong: A Randomised Controlled Trial
Brief Title: Promoting Adolescent Development Through Sports in Hong Kong
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Sports2013HK
Record Dates: First submitted 2013-09-27; First posted 2013-10-07 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Adolescent Development
Keywords: Positive youth development; Sports / physical activity
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Health Promotion

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sports mentorship programme (Experimental): 1.5-hour sports mentorship session once a week, 18 weeks total.
  Interventions: Behavioral: Sports mentorship programme
- Health promotion (Active Comparator): The access to a health promotion website any time during the intervention period. The website contains general health information including those related to physical activity.
  Interventions: Behavioral: Health promotion

INTERVENTIONS:
Behavioral: Sports mentorship programme — 1.5-hour sports mentorship session once a week, 18 weeks total.
  Other Names: Physical activity; Sports
  Arms: Sports mentorship programme
Behavioral: Health promotion — The access to a health promotion website any time during the intervention period. The website contains general health information including those related to physical activity.
  Arms: Health promotion

SUMMARY:
Background

A physically active lifestyle is crucial for development but a large number of youth in Hong Kong are sedentary and do not meet the International (World Health Organisation) and the local (Leisure and Cultural Services Department) recommendation for physical activity. On the other hand, the evidence for implementing positive youth development programme through physical activity and sports is elusive.

Purpose

This study aimed to promote physical activity and sports amongst adolescents in Hong Kong through a structured sports mentorship intervention. The study also aimed to investigate the effect of such programme in positive youth development.

Methods

This was a two-phased study with Phase I being the preparatory stage and Phase II being the implementation stage. In Phase I, questionnaire surveys and focus group interviews were conducted to understand the relevant perceptions and opinions amongst various stakeholders (e.g. teachers, parents, and students). The data collected was analysed to inform the design and planning of the Phase II intervention. Phase II was an experimental trial of our sports mentorship programme. Participating students were divided into intervention and control group, where the former received the sports mentorship programme and the later did not. The intervention was 18 weeks long providing an additional 90 minutes of active time per week for all students in the intervention group. Programme mentors were trained and supported in reference to previous evidence. Intervention effectiveness were evaluated by comparing the outcomes between intervention and control group.

DETAILED DESCRIPTION:
Introduction

Physical activity is beneficial to all aspects of health, from physical fitness and metabolic control to mental and psychosocial well-being. These benefits are particularly important to children and adolescents as they are undergoing an active development and building up a foundation for their future success. Unfortunately, Hong Kong children are becoming less and less physically active. Data from government surveys in 2009 showed that only 34.2% of children aged 7 to 12 years had at least 60 minutes of moderate or vigorous activity five days a week over a 3 month period. Another recent survey reported that only 6.6% of secondary school students in Hong Kong met the WHO recommended standard of physical activity - 60 minutes of moderate and vigorous activity every day. In fact, 27.1% of adolescents did not even have moderate and vigorous physical activity in any days of the past week.

Upsurging adolescent problems have been identified in Hong Kong, including smoking, underage drinking, substance abuse, and the deterioration of mental well-being (D. T. Shek, 2006). Take mental health as an example. Mental health problems were estimated to affect 10 to 20% of children and adolescents worldwide (Kieling et al., 2011), resulting in short-term and long-term adverse consequences (Johnson, Roth, Schultz, & Breslau, 2006). Conventionally, mental health problems were tackled using a disease model, which focuses on disease treatment. However, it has been more recognised in recent decade that primary prevention would be important to improve the overall mental well-being of children and adolescents (Kieling et al., 2011).

Instead of the traditional disease model, strength-based positive prevention models has been called upon, where Positive Youth Development (PYDs) is one of the most successful one targeting adolescents. To understand the concept of PYD, it is important to have a glimpse at the traditional view of adolescence. The transition period located at the second decade of the human lifespan was conventionally regarded as the period of 'storm and stress' (Hall, 1904). It was suggested that adolescents often alternate between the extremes of sorrow and exuberance (N. Holt, 2008). Nonetheless, it was later recognised that the emphasis on these negative characteristics was disproportionately too much and a new perspective on adolescent development emerged. This new perspective is later named the PYD. Instead of the conventional deficit-reduction (or 'disease') approach, the PYD focuses on how to strengthen adolescents' internal and external asset so that problems could be prevented or alleviated. Since the establishment of this new concept in the 80s and 90s, a growing number of research has been conducted to investigate the actual implementation of such model.

The PYD model could be implemented in many context, but it is argued that sports and physical activity is one of the most suitable (Fraser-Thomas, Cote, & Deakin, 2005; Larson, 2000; Perkins & Noam, 2007). Actually such claim was consistent with the 'QK Blog', an existing adolescent strengthening platform (Kwai Tsing Safe Community and Healthy City Association, 2012). Nevertheless, the actual benefit of these sports-based PYD problem was rarely investigated, especially in China (Coakley, 2011; Fraser-Thomas et al., 2005). Therefore, we conducted the present project to promote two major aspects among adolescents in Hong Kong: physically activity and adolescent development.

Purpose/Objectives/Aims

This project will explore the possibility of fostering positive adolescent development through tailoring a community-based youth project in Kwai Tsing district in Hong Kong. Specifically, physical activity would benefit the adolescents in terms of physical, psychological/emotional, and social development, together of which forms the important foundation for a healthy and productive adult life. The project will incorporate a physical activity intervention guided by behavioural theory in a secondary school-based setting.

Project

Overview

This is a two-phase project with Phase I being the preparatory stage and Phase II being the Implementation stage. Phase I mainly focused on the attitude, perceived benefits and barriers among various stakeholders, including students, parents, and teachers. The stakeholders were then interviewed in a focus group setting or surveyed using questionnaires.

The data collected in Phase I were then analysed, which guided the design and implementation of Phase II - the actual implementation of the intervention. In addition to the results of Phase I, a thorough literature search were also conducted in order to understand the existing evidence regarding the correlates of physical activity as well as the theoretical construct in promoting adolescent development through sports / physical activity.

Recruitment

To ensure sufficient support from the school, we contacted the secondary schools with physical education teacher graduated from the Department of Physical Education, Hong Kong Baptist University. A formal invitation letter were sent to each school, outlining the background, implementations, and expected outcomes of the programmes. Telephone calls were also made to each schools' principal, extra-curricular master, or physical education (PE) panel heads for discussing the feasibility and other details of implementing the programme in their school. To allow flexibility, schools may only participate in either Phase I or Phase II or both, depending on their preference.

The Phase I PE teacher survey questionnaires were sent directly to all the 454 secondary schools. All schools in Hong Kong were invited so as to obtain a more representative sample, which may inform both the current intervention programme and relevant research and services in the future.

Intervention Design

Design of the intervention was guided by both the empirically results of Phase I and a through literature review. The theoretical framework and the practical implementation of the interventions are as follows:

Framework

Our programme was informed by two theoretical frameworks: first, the Theory of Planned Behaviour (TPB) for encouraging students' participation in sports and PA, and second, the Positive Youth Development (PYD) framework for enhancing students' holistic development.

The TBP is a successful framework in predicting physical activity behaviour in young people (Craig, Goldberg, & Dietz, 1996). It was found that attitude, perceived behavioural control, and subjective social norm has a strong influence in taking part physical activity. In particular, the effect of self-efficacy and attitude on PA were even significant after controlling for youth's past PA habit. In other words, improving students' self-efficacy and attitude may increase their participation in PA, regardless of their current activity level.

Whereas the TBP could assist in motivating students' participation in PA, the PYD framework may help to define the structure of the programme for enhancing holistic adolescent development. Specifically, we adapted the United States National Research Council and Institute of Medicine (NRCIM) suggestion in developing this programme.

Apart from these principles, we also blended in well-established psychological theories in the present programme. For example, we regarded the person who guide and facilitate the exercise sessions to be 'mentors' instead of 'coaches'. These mentors did not only teach students sporting skills, but were also responsible to maintain the exercise sessions fun, democratic and empowering. The mentors were also educated with the means in establishing a 'mastery-oriented' atmosphere, instead of a 'performance-oriented' one, during teaching and exercising. The former attitude encourages a constant improvement for each of the students while the later one encourages comparison of performance within the group. Previous psychological experiments have shown that people in mastery-oriented attitude would be more motivated in constant improvements. All the mentors of the programme were introduced with the present programme principle and supported by our project members, including health and physical education experts.

Implementation

Eighteen 1.5-hour activity sessions were carried out weekly for all students participating in this programme. The total activity time for each student was 27 hours. The quantity 1.5 hours per week was chosen to conform the physical activity baseline indicator of the Hong Kong Leisure and Cultural Services Department (Department of Sports Science & Physical Education of The Chinese University of Hong Kong, 2009).

Roughly speaking, the programme could be categorised into four stages: Introduction / Recapitulation, Goal Setting, Skill Building, and Reflection. The Introduction / Recapitulation stages were for students and mentors to warm up and building their bonds. Mentors were advised to set up their own rules with students within these periods. Exercises and physical activities during these sessions were designed to be relatively easy for encouragement and motivation purpose. The Goal Setting stages were transition periods where students were assisted in establishing their own goals during the programme. During these stages, mentors helped students in realising their current sporting skills, which acted as the starting point of goal setting. Skill Building stages were the major components of the programme. Students were instructed to reach their own goals through practice and play. Finally, the Reflection sessions were for students reflect on their own improvement and barriers encountered during the Skill Building stages with the assistance of the mentors. The inclusion of reflections ensured that students' benefits in the programme were consolidated and could be sustained in a longer period. Details of the intervention frameworks, principles, implementations, and mentor education could be found in the Programme Guidebook for Mentors)

ELIGIBILITY:
Inclusion Criteria:

* Form 1 and 2 students in the 12 participating schools.

Exclusion Criteria:

* Students who cannot comprehend Cantonese
* Students who are physically unfit for school physical education lessons

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 719 (Actual)
Dates: Start 2013-09; Primary Completion 2014-07 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Psychological development | One-month after intervention
  Mental Component Summary score (MCS-12) of the Chinese (HK) SF-12v2 Health Survey. General Self-efficacy Scale and Connor-Davidson Resilience Scale

SECONDARY OUTCOMES:
Social development | One-month after intervention
  Resnick School and Family Connectedness Scales and perceived social support.
Sleep quality | One-month after intervention
  Pittsburgh Sleep Quality Index
Obesity status | One-month after intervention
  IOTF body-mass-index and bioimpedance method
Physical fitness | One-month after intervention
  Physical fitness would be measured by physical fitness test comprising of standing long jump, sit-and-reach, and sit-ups.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Ip, Dr., Principal Investigator — The University of Hong Kong
Locations (1):
- University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided